CLINICAL TRIAL: NCT02477371
Title: Fractional Flow Reserve Versus Angiography Randomization for Graft Optimization Trial
Acronym: FARGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anne Langhoff Thuesen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20130050
Record Dates: First submitted 2015-01-19; First posted 2015-06-22 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Arteriosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fractional flow reserve-guided CABG (Experimental): Patients are randomized to an FFR-guided CABG. FFR-measurements are made on coronary arteries with intermediate stenoses, that are planned for grafting. The FFR-values are blinded for both the operator, the patient and the heart team meeting. The graft plan form the heart team meeting are changed by the study investigator according to the FFR-measurements and randomization, so that coronary arteries with FFR ≤ 0,8 receive grafting and coronary arteries with FFR > 0,8 are deferred.
  Interventions: Procedure: Fractional flow reserve-guided CABG
- Angiography-guided CABG (Active Comparator): Patients are randomized to an angiography-guided CABG. FFR-measurements are made on coronary arteries with intermediate stenoses, that are planned for grafting. The FFR-values are blinded for both the operator, the patient and the heart team meeting. The graft plan are based on the coronary angiography.
  Interventions: Procedure: Angiography-guided CABG

INTERVENTIONS:
Procedure: Fractional flow reserve-guided CABG — Coronary arteries with angiographical significant stenoses, that are planned for grafting at the heart team meeting and where FFR-measurements are made, only receive grafting if FFR-value is ≤ 0,8. Arteries with FFR-values > 0,8 are deferred.
  Arms: Fractional flow reserve-guided CABG
Procedure: Angiography-guided CABG — Coronary arteries with angiographical significant stenoses, that are planned for grafting at the heart team meeting all receive grafting. FFR-measurements are still made, but not used for guidance of grafting.
  Arms: Angiography-guided CABG

SUMMARY:
The FARGO trial is a prospective, randomized (1:1), multicenter study. The aim of the study is to assess the importance of fractional flow reserve (FFR) assessment prior to coronary artery bypass grafting (CABG) with respect to planning and guiding the revascularization strategy. The study compares an FFR-guided strategy to an angiography-guided strategy in patients planned for surgical revascularization.

DETAILED DESCRIPTION:
FFR measurements are made on all patients that enters the study. FFR measurements on coronary arteries with intermediate stenoses, that are planned for grafting, are done before CABG is performed. Patients are randomized to either an FFR-guided CABG or an Angiography guided CABG.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina or unstable angina / NSTEMI (Non ST segment elevation myocardial infarction) candidate to CABG
* At least one study lesion, which is an intermediate lesion planned for grafting at the Heart Team Meeting.(Definition of Study lesions: ≥ 50% stenosis of a major epicardiel artery (where the proximal reference segment has a diameter> 2.5 mm), which can be passed with a FFR-wire without significant risk. Study Lesions can be drawn from all coronary arteries.)
* Signed informed consent form

Exclusion Criteria:

* Significant valvular disease with indication to surgical treatment
* Previous open-heart-surgery
* Left main lesion without other intermediate lesions
* Treatment with Persantin Retard
* One vessel disease
* Renal impairment (creatinine ≥ 150 umol / l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage open grafts of all grafts | 6 months
  Open graft definition: graft with TIMI III flow with no anastomosis stenosis (TIMI flow grades based on results of the Thrombolysis In Myocardial Infarction trial)

SECONDARY OUTCOMES:
Graft stenosis (shaft and anastomoses) | 6 months
Change in CCS class from index to follow-up (FU) | 6 months
  CCS class (Canadian Cardiovascular Society grading of angina)
Change in Quality of life (EQ-5D) from index to FU | 6 months
MACCE (Major Adverse Cardiac and Cerebrovascular event: death, myocardial infarction, stroke, new revascularization by CABG or PCI (Percutaneous coronary intervention) | 6 months
Procedural maximum Troponin I (cTnI), Troponin T (TnT) or creatinine kinase MB (CKMB) values depending on local conditions. | The first 24 hours after the operation
Procedure time | During surgery (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Langhoff Thuesen, MD, Principal Investigator — Department of Cardio-thoracic surgery, Odense University Hospital; Lisette Okkels Jensen, MD,PhD,DMSc, Study Director — Department of Cardiology, Odense University Hospital; Per Thayssen, MD, DMSc, Study Chair — Department of Cardiology, Odense University Hospital; Poul Erik Mortensen, MD, Study Chair — Department of Cardio-thoracic surgery, Odense University Hospital
Locations (3):
- Denmark (3):
  - Department of Cardiology and Cardiothoracic surgery, Aarhus University Hospital, Skejby Sygehus, Aarhus, Aarhus N
  - Anne Langhoff Thuesen, Odense, Odense C
  - Department of Cardiology and Cardiothoracic surgery, Aalborg University Hospital, Aalborg

REFERENCES:
- [Derived] Thuesen AL, Riber LP, Veien KT, Christiansen EH, Jensen SE, Modrau I, Andreasen JJ, Borregaard B, Junker A, Mortensen PE, Jensen LO. Health-Related Quality of Life and Angina in Fractional Flow Reserve- Versus Angiography-Guided Coronary Artery Bypass Grafting: FARGO Trial (Fractional Flow Reserve Versus Angiography Randomization for Graft Optimization). Circ Cardiovasc Qual Outcomes. 2021 Jun;14(6):e007302. doi: 10.1161/CIRCOUTCOMES.120.007302. Epub 2021 Jun 3. PMID 34078097
- [Derived] Thuesen AL, Riber LP, Veien KT, Christiansen EH, Jensen SE, Modrau I, Andreasen JJ, Junker A, Mortensen PE, Jensen LO. Fractional Flow Reserve Versus Angiographically-Guided Coronary Artery Bypass Grafting. J Am Coll Cardiol. 2018 Dec 4;72(22):2732-2743. doi: 10.1016/j.jacc.2018.09.043. PMID 30497559